CLINICAL TRIAL: NCT06911853
Title: Enhancing Clinical and Cultural Virtual Encounter in Health Professional Students: 3 Is (Internationalization, Innovation, Interdisciplinary) in Action
Acronym: 3I in action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chan Siu Ling, Senior Lecturer of School of Nursing, Principal Investigator, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HKWC-2022-389; 899 (Other Grant/Funding Number: HKU)
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Interprofessional Education
Keywords: Interprofessional education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Reality Group (Experimental)
  Interventions: Other: Virtual Reality Videos

INTERVENTIONS:
Other: Virtual Reality Videos — Based on the Phase of Engagement Framework, two online orthopaedic modules focusing on interprofessional and intercultural educations on low back pain (LBP) and adolescent idiopathic scoliosis (AIS) were developed. The students (n=104) were randomized into two groups. In the first module, the Virtual Reality Group as the intervention group received a virtual reality (VR)-enhanced LBP education, while the Case-based Learning Group as the control group engaged with a case study on LBP. After a 3-week washout period, the groups crossed over: the the Virtual Reality Group as the intervention group received the VR-enhanced education on AIS, and the Case-based Learning Group as the control group focused on an AIS case study.

SUMMARY:
This is a cross-over randomized control study with 3 time-points' measurement. This study is mainly to evaluate if the online pedagogic innovative learning modules could benefit students through their interprofessional and intercultural virtual encounters, with a focus on assessing their cultural awareness, interprofessional attitude and online learning engagement.

DETAILED DESCRIPTION:
This study aims to promote and implement internationalization, innovative and intedisciplinary teaching and learning strategies through the set up of online modules of selected topics of interest. The specific objectives are: :

To enhance the educational outcomes of students from respective health disciplines in interdisciplinary learning via case-based clinical scenarios adopted in the online modules; To develop internationalization experience among students of different countries in terms of intercultural learning through the cultural exchange; To assess level of students' empowerment in active learning via 'student-as-partner' initiatives in the cultural exchange; To evaluate the effectiveness of online learning engagement among students through participating in the online modules.

Based on the Phase of Engagement Framework, two online orthopaedic modules focusing on interprofessional and intercultural educations on low back pain (LBP) and adolescent idiopathic scoliosis (AIS) are developed. The students (n=104) are randomized into two groups using SNOSE. In the first module, one group receives a virtual reality (VR)-enhanced LBP education (intervention group), while the other group engages with a case study on LBP (control group). After a 3-week washout period, the groups cross over: the intervention group receives the VR-enhanced education on AIS, and the control group focuses on an AIS case study. Interprofessional learning experience, cultural awareness, and online learning engagement are measured using validated tools at three time points (baseline, after first and second modules).

ELIGIBILITY:
Inclusion Criteria:

* undergraduate healthcare students

Exclusion Criteria:

* cannot communicate in English

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Both gender are welcomed to participate in the study
Enrollment: 104 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Students' Perceptions of Interprofessional Clinical education - Revised | 2 months
  Using Students' Perceptions of Interprofessional Clinical Education-Revised (SPICE-R) as the tool to measure the increased level of interprofessional learning experiences. The SPICE-R instrument includes ten items, and is divided into three factors: interprofessional teamwork and team-based practice (items 1, 5, 6, 8, 9 and 10), roles/responsibilities for collaborative practice (items 2 and 7), and patient outcomes from collaborative practice (items 3 and 4). It is a 5-point Likert scales (1 = 'strongly disagree' and 5 = 'strongly agree') with score ranging from 10-50. SPICE-R was chosen for its strong psychometric properties including reliability and construct validity (Dominguez et al., 2016; Lockeman et al., 2017). The instrument has high composite reliability at 0.84, indicating strong validity based on established criteria. Higher score on SPICE-R reflect more positive interprofessional experiences.

CONTACTS AND LOCATIONS:
Locations (1):
- 5/F, Academic Building, 3 Sassoon Road, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No